CLINICAL TRIAL: NCT04700189
Title: A First in Human Clinical Trial to Evaluate the Safety and Effectiveness of the STREAMLINE™ SURGICAL SYSTEM in Patients With Open-Angle Glaucoma
Brief Title: A FIH Trial of the STREAMLINE™ SURGICAL SYSTEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New World Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DF6-CL-20-03
Record Dates: First submitted 2020-12-18; First posted 2021-01-07 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Intraocular Pressure; Open Angle Glaucoma
Keywords: Intraocular Pressure; Glaucoma; Glaucoma Surgery; Ab interno
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment with Streamline following cataract surgery (Experimental): Treatment with Streamline System following phacoemulsification
  Interventions: Device: ab interno canaloplasty

INTERVENTIONS:
Device: ab interno canaloplasty — A modification of traditional canaloplasty procedure. Can be combined with or done without cataract surgery.

SUMMARY:
The purpose of this study is to evaluate the safety and Intraocular pressure lowering effectiveness of the Streamline™ Surgical System.

DETAILED DESCRIPTION:
This is a prospective, nonrandomized, open-label study evaluating the safety and IOP-lowering effectiveness of CPI Visco-Surgical System (STREAMLINE™ SURGICAL SYSTEM) in patients with open-angle glaucoma undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria in order to be eligible for participation in this study:

1. Subjects qualifying for cataract surgery
2. Subjects with diagnosis of open-angle glaucoma in at least one eye with unmedicated IOP of 21-36 mmHg.

Exclusion Criteria:

* Subjects are ineligible for participation in this study if s/he meets any of the following criteria:

  1. Patients who could not be washed-out of IOP-lowering medications. .

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Proportion of unmedicated eyes with intraocular pressure (IOP) reduction of ≥20% | From Baseline at Month 12
  Descriptive

SECONDARY OUTCOMES:
Changes from baseline in intraocular pressure (IOP) | From Baseline at Month 12
  Exploratory analysis
Changes from baseline in number of IOP lowering medications | From Baseline at Month 12
  Exploratory analysis

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Lozcano, MD, Principal Investigator — Puebla, Mexico
Locations (1):
- Dr. Gabriel S. Lazcano Gomez, Puerto México, Mexico